CLINICAL TRIAL: NCT02512939
Title: Predictive Values of Next Generation Interferon Gamma Release Assays for Latent Tuberculosis Infection
Acronym: NextGen
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University College, London (Other)
Collaborators: Public Health England (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Next gen
Record Dates: First submitted 2015-07-28; First posted 2015-07-31 (Estimated); Last update posted 2023-05-16 (Actual); Status verified 2023-05

CONDITIONS: Tuberculosis
Keywords: tuberculosis; diagnostic test
MeSH Terms: conditions — Tuberculosis | interventions — Hematologic Tests

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Contacts of TB cases (Experimental): Blood test, not yet marketed, development phase
  Interventions: Procedure: blood test, not yet marketed, no trade name

INTERVENTIONS:
Procedure: blood test, not yet marketed, no trade name — blood test using the new TB diagnostic test

SUMMARY:
This study will assess the next generation of blood tests for latent TB infection, which may be able to indicate how treatment is working as well as in diagnosis infection.

DETAILED DESCRIPTION:
Currently available blood tests for latent tuberculosis infection (LTBI) identify people who have been previously infected with M. tuberculosis. Whilst they are sensitive and specific, they cannot be used to monitor the effectiveness of treatment for LTBI. New blood tests ("fourth generation Quantiferon tests") give a more complete measurement of the workings of the immune system, which may be useful to show whether treatment is working. These new tests have not yet been evaluated in clinical practice, so their usefulness in identifying people at highest risk of TB disease and monitoring treatment is unknown.

Mass gatherings, such as the annual Hajj pilgrimage, may encourage the spread of infectious diseases, including respiratory infections such as influenza, respiratory syncytial virus, and possibly also tuberculosis. However, the risk of TB infection during the Hajj has not been reliably measured. It is important to measure this risk so that pilgrims can be given suitable advice about preventing infection.

ELIGIBILITY:
Inclusion Criteria:

- Contacts: Adult (aged 16 years or older) contacts of smearpositive pulmonary TB patients attending participating TB clinics or primary care centres for screening will be invited to take part. Contacts will include all individuals with a cumulative duration of exposure of greater than eight hours to the relevant index case in a confined space during the period of infectiousness (prior to initiation of treatment). Patients with active TB: Newly diagnosed, microbiologically confirmed tuberculosis disease (pulmonary or extrapulmonary) attending participating TB clinics or primary care centres. Hajj pilgrims: Individuals arranging travel to Saudi Arabia for the Hajj through participating tour operators.

Exclusion Criteria:

- Contacts: Active TB disease. Individuals who are unable to give informed consent. Children aged under 16 years.

TB cases: Individuals who are unable to give informed consent. Children aged under 16 years.

Hajj pilgrims: Active TB disease. Any health indication which would prevent travel to Saudi Arabia. Individuals who are unable to give informed consent. Children aged under 16 years.

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 675 (Actual)
Dates: Start 2015-07; Primary Completion 2016-11-30 (Actual); Study Completion 2016-11-30 (Actual)

PRIMARY OUTCOMES:
assess prognostic ability of blood test by assessing development of active TB disease compared to the current gold standard | 1 year
  assess prognostic ability of blood test by assessing development of active TB disease.

SECONDARY OUTCOMES:
assess the sensitivity of new blood tests for detecting TB infection in patients with active TB disease compared to teh current godl standard | 1 year
  estimate the sensitivity of new blood tests for detecting TB infection in patients with active TB disease
estimate the risk of infection with M. tuberculosis and other respiratory pathogens amongst UK pilgrims undertaking the Hajj. | 1 year
  estimate the risk of infection with M. tuberculosis and other respiratory pathogens amongst UK pilgrims undertaking the Hajj.

CONTACTS AND LOCATIONS:
Overall Officials: Ibrahim Abubakar, PhD, Principal Investigator — University College, London
Locations (5):
- United Kingdom (5):
  - Barts NHS Trust, London
  - Ealing Hospital, London
  - North Middlesex Hospital, London
  - Northwick Park Hospital, London
  - West Middlesex Hospital NHS Trust, London

IPD SHARING:
Plan to Share IPD: No